CLINICAL TRIAL: NCT01109641
Title: PhrenIc Nerve mappinG and Stimulation EP Catheter Study: PING-EP Study
Acronym: PING-EP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Italia (Industry)
Responsible Party: Francesco De Seta, Medtronic Italia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT-PINGEP
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: diagnostic electrophysiology catheter — electrical measurements through a diagnostic electrophysiology catheter

SUMMARY:
The PING-EP study is designed to evaluate electrode properties on phrenic nerve stimulation (PNS) in coronary sinus using a commercially available diagnostic electrophysiology catheter.

ELIGIBILITY:
Inclusion Criteria:

* Subject is indicated for a cardiac resynchronization therapy-pacemaker or defibrillator (CRT-P/CRT-D) implant, for an upgrading from a previously implanted single/dual chamber pacemaker/implantable cardioverter (ICD) or for system revision requiring repositioning of the transvenous left ventricular (LV) lead
* Patient has signed and dated the study-specific Patient Informed Consent form
* Subject is at least 18 years of age

Exclusion Criteria:

* Patient has a previous LV lead implanted not requiring repositioning
* Pregnant woman
* Patient is enrolled or planning to participate in any concurrent study, which would confound the results of this trial as determined by Medtronic, during the course of this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Effect of electrode property on phrenic nerve stimulation (PNS) | at implant
  Effect of electrode property on PNS in the cardiac veins

SECONDARY OUTCOMES:
Effect of electrode configuration on phrenic nerve stimulation (PNS) | at implant
Electrode polarity effect on phrenic nerve stimulation (PNS) | at implant
Effect of electrode property on sensing (r-wave amplitude) | at implant
Incidence of phrenic nerve stimulation (PNS) in the cardiac veins | at implant
  Incidence of PNS occurrence in different locations in the cardiac vein

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Biffi, Principal Investigator — Policlinico S. Orsola Malpighi, Bologna, Italy; Francesco Zanon, Principal Investigator — Ospedale S. Maria della Misericordia, Rovigo, Italy; Luigi Padeletti, Principal Investigator — Azienda ospedaliero-universitaria Careggi, Firenze, Italy; Manuel Bertaglia, Principal Investigator — Azienda Unità Socio Sanitaria di Dolo Mirano, Mirano (VE), Italy
Locations (4):
- Italy (4):
  - Azienda Ospedaliero-Universitana di Bologna, Policlinico S. Orsola Malpighi, Bologna, Bologna
  - Azienda Ospedaliero-universitaria Careggi, Florence, Firenze
  - Ospedale S. Maria della Misericordia, Rovigo, Rovigo
  - Azienda Unità Socio Sanitaria di Dolo Mirano, Mirano, Venezia

REFERENCES:
- [Background] McAlister FA, Ezekowitz J, Hooton N, Vandermeer B, Spooner C, Dryden DM, Page RL, Hlatky MA, Rowe BH. Cardiac resynchronization therapy for patients with left ventricular systolic dysfunction: a systematic review. JAMA. 2007 Jun 13;297(22):2502-14. doi: 10.1001/jama.297.22.2502. PMID 17565085
- [Background] Gurevitz O, Nof E, Carasso S, Luria D, Bar-Lev D, Tanami N, Eldar M, Glikson M. Programmable multiple pacing configurations help to overcome high left ventricular pacing thresholds and avoid phrenic nerve stimulation. Pacing Clin Electrophysiol. 2005 Dec;28(12):1255-9. doi: 10.1111/j.1540-8159.2005.00265.x. PMID 16403156
- [Background] Albertsen AE, Nielsen JC, Pedersen AK, Hansen PS, Jensen HK, Mortensen PT. Left ventricular lead performance in cardiac resynchronization therapy: impact of lead localization and complications. Pacing Clin Electrophysiol. 2005 Jun;28(6):483-8. doi: 10.1111/j.1540-8159.2005.40066.x. PMID 15955178
- [Background] Alonso C, Leclercq C, d'Allonnes FR, Pavin D, Victor F, Mabo P, Daubert JC. Six year experience of transvenous left ventricular lead implantation for permanent biventricular pacing in patients with advanced heart failure: technical aspects. Heart. 2001 Oct;86(4):405-10. doi: 10.1136/heart.86.4.405. PMID 11559679
- [Background] Knight BP, Desai A, Coman J, Faddis M, Yong P. Long-term retention of cardiac resynchronization therapy. J Am Coll Cardiol. 2004 Jul 7;44(1):72-7. doi: 10.1016/j.jacc.2004.03.054. PMID 15234410
- [Background] Ellery S, Paul V, Prenner G, Tscheliessnigg K, Merkely B, Malinowski K, Frohlig G, Hintringer F, Bosse O, Diotallevi P, Ravazzi AP, Flathmann H, Danilovic D, Unterberg-Buchwald C; OVID Study Investigators. A new endocardial "over-the-wire" or stylet-driven left ventricular lead: first clinical experience. Pacing Clin Electrophysiol. 2005 Jan;28 Suppl 1:S31-5. doi: 10.1111/j.1540-8159.2005.00084.x. PMID 15683519
- [Background] Matsumoto Y, Krishnan S, Fowler SJ, Saremi F, Kondo T, Ahsan C, Narula J, Gurudevan S. Detection of phrenic nerves and their relation to cardiac anatomy using 64-slice multidetector computed tomography. Am J Cardiol. 2007 Jul 1;100(1):133-7. doi: 10.1016/j.amjcard.2007.01.072. Epub 2007 May 21. PMID 17599455